CLINICAL TRIAL: NCT04795856
Title: Understanding the Metabolic and Functional Derangement of Primary Mitral Regurgitation: a Feasibility Study Using C-11 Acetate Cardiac PET-MRI
Brief Title: Understanding the Metabolic and Functional Derangement of Primary Mitral Regurgitation: a Feasibility Study Using Carbon 11(C-11) Acetate Cardiac Positron Emission Tomography Magnetic Resonance Imaging (PET-MRI)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of recruitment and PI departure
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pradeep Bhambhvani, MD, Professor, Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R20-178
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — carbon-11 acetate

STUDY DESIGN:
Intervention Model Description: The healthy group will establish a baseline for the moderate- severe mitral valve regurgitation (PMR) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- chronic compensated moderate-severe primary mitral regurgitation (PMR) (Active Comparator)
  Interventions: Drug: [11C] acetate
- Healthy Volunteers (Active Comparator)
  Interventions: Drug: [11C] acetate

INTERVENTIONS:
Drug: [11C] acetate — PET Tracer

SUMMARY:
The aim of this pilot imaging study is to investigate the underlying changes in myocardial oxidative metabolism, myocardial inflammation and alterations in extracellular volume in patients with chronic compensated moderate-severe primary mitral regurgitation (PMR). The PET tracer [11C] acetate will be used to image and quantify myocardial oxygen consumption (MVO2) in hearts of the study participants. Cardiac magnetic resonance imaging (CMR) using a gadolinium-based contrast agent (GBCA) will be performed to assess for and quantify expansion of myocardial extracellular volume (ECV) and myocardial inflammation. We will enroll a total of 12 participants, nine of whom will be patients with chronic, compensated asymptomatic moderate-severe PMR evaluated at the UAB Cardiovascular Disease and Structural Valve Clinic and three normal control subjects.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Patients with chronic, asymptomatic, compensated PMR evaluated in the UAB Structural Valve Clinic OR Normal controls identified from a normal aged matched population.
* Negative urine or serum β-human chorionic gonadotropin (hcg) test within 48 hours of [11C] acetate administration in women of childbearing potential. Women who are post-menopausal with at least 1 year since last menses or documented surgical sterilization will not require pregnancy testing.

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Inability to lie still for the imaging study
* Weight exceeding the weight limit of the PET imaging table (500 pounds)
* Comorbidities including any of the following: history of coronary artery disease, prior coronary revascularization, prior myocardial infarction, prior open sternotomy, history of congestive heart failure, history of non-ischemic cardiomyopathy including dilated, restrictive, hypertrophic, amyloid heart disease, cardiac sarcoidosis, history of hypertension, diabetes mellitus, chronic kidney disease with a glomerular filtration rate (GFR) less than 60 ml/min/1.73 m2 , history of other valvular heart disease defined as mitral stenosis, aortic stenosis, more than mild aortic regurgitation, more than mild tricuspid regurgitation, history of more than mild pulmonary hypertension and history of cancer with exposure to chemotherapy or radiotherapy.
* Contraindication for gadolinium-based contrast agent, ProHance (gadoteridol)
* Contraindication for MRI study (e.g. non-removable metal implants or certain tattoos)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-06 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Quantitatively correlate metabolic findings from the PET component with quantitative T1 and T2 parametric mapping from the cardiac MR component of the hybrid PET-MR study. | 0-48 hours
  Parametric analysis of T1 and T2 mapping will be performed using dedicated software (Qmap, Medis).

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhambhvani, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No